CLINICAL TRIAL: NCT06427876
Title: FASENRA® Subcutaneous Injection 30 mg / 10mg Syringe Protocol of Specific Drug Use Result Study for Pediatric Patients
Brief Title: Fasenra Pediatric Japan Post-Marketing Study(PMS)
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250C00100
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
The purpose of the investigation is to confirm the followings under the post-marketing actual use of Fasenra® Subcutaneous Injection 30 mg / 10mg Syringe (hereinafter referred to as Fasenra).

1. Development of unexpected related AEs*
2. To grasp development of related AEs* in the real-world post-marketing setting.
3. Effectiveness (pulmonary function and asthma control) * AEs investigator or MAH considers that there is a reasonable possibility that the experience may have been caused by the drug

DETAILED DESCRIPTION:
This investigation will be conducted to support the application for re-examination specified in Article 14-4 of the Act on Securing Quality, Effectiveness and Safety of Products Including Pharmaceuticals and Medical Devices.

The purpose of the investigation is to confirm the followings under the post-marketing actual use of Fasenra® Subcutaneous Injection 30 mg / 10mg Syringe (hereinafter referred to as Fasenra).

1. Development of unexpected related AEs*
2. To grasp development of related AEs* in the real-world post-marketing setting.
3. Effectiveness (pulmonary function and asthma control) * AEs investigator or MAH considers that there is a reasonable possibility that the experience may have been caused by the drug

ELIGIBILITY:
Inclusion Criteria:

The evaluable patients in children aged ≥6 years to <15 years are those treated with Fasenra for the first time due to "Bronchial asthma (only the patients with intractable bronchial asthma which could not be controlled with the existing therapy)

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The evaluable patients in children aged ≥6 years to <15 years are those treated with Fasenra for the first time due to "Bronchial asthma (only the patients with intractable bronchial asthma which could not be controlled with the existing therapy)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADRs | from baseline to 1year
  The incidence of ADRs related to Fasenra Safety Specification, Serious infection and other

CONTACTS AND LOCATIONS:
Overall Officials: Shunsuke Hiroki, Study Director — AstraZeneca
Locations (10):
- Japan (10):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Mie
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home